CLINICAL TRIAL: NCT05347875
Title: Exploring the Influence of a Novel Application for Training and Evaluating Walking Implementation of an App-based Walking Aid Skills Training Program Aid Skills in Walking Aid Users: A Protocol for a Pragmatic Single-blind Randomized Controlled Trial
Brief Title: Implementation of an App-based Walking Aid Skills Training Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); Laval University (Other); CIRISS (Unknown)
Responsible Party: Principal Investigator, Ranita Manocha, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB21-1165
Record Dates: First submitted 2022-04-14; First posted 2022-04-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lower Limb; Sprain (Strain); Lower Limb Fracture; Stroke; Multiple Sclerosis
Keywords: Gait aid; Walking aid; Cane; Crutch; Walker
MeSH Terms: conditions — Sprains and Strains; Stroke; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Breathing Skills App
  Interventions: Other: Breathing skills app
- Experimental Group (Experimental): ICanWALK© App
  Interventions: Other: Walking aid skills app

INTERVENTIONS:
Other: Walking aid skills app — The interventional app teaches users how to fit, walk with, and navigate stairs and chairs with a walking aid. It contains instructional videos with key "components" of these skills highlighted. The user can use their phone's video to record themselves performing the taught skills to enable them to review their usage of the walking aids.
  Other Names: ICanWALK
  Arms: Experimental Group
Other: Breathing skills app — This app has the same interface as the ICanWALK app. Instead, it teaches deep breathing for stress relief and breathing to improve lung function.
  Arms: Control Group

SUMMARY:
Walking aids (WA), such as crutches, canes, and walkers allow individuals to move independently after lower body impairment. Improper WA use may lead to upper body discomfort, pain, or injury. Improper WA use has been associated with increased risk of falls, which may result in traumatic brain injury or even death. WA-related accidents and injuries may not only affect an individual patient's quality of life; they may also increase healthcare system resource use and caregiver burden. WA-related injuries may be preventable if WA are properly fit and sufficient training is provided to the WA user.

Smartphone applications (apps) are widely used technologies that have been used to improve health outcomes in populations of healthy and chronically ill individuals. We have developed an app that can be used to teach WA users how to properly fit and use their devices. This app is called Improving Canadians' Walking Aid skills, Learning, and Knowledge (ICanWALK©).

The development of the Walking Aids Skills Test© (WAST©) allows for the objective measurement of how well an individual uses their walking aid. It is important to develop such a measurement in order to see whether interventions such as mobile applications change a walking aid user's ability to walk with their device. This 12-item objective evaluation measures the ability of an individual to use their walking aid in different settings, while picking up an object off the ground, navigating stairs, or encountering terrains such as gravel or grass.

Three hypotheses will be explored through this clinical trial. Hypothesis 1: Patients who use the ICanWALK© app will have improved balance confidence compared to the control group.

Hypothesis 2: Patients who use the ICanWALK© app will have improved balance, improved mobility, less pain, and fewer falls compared to the control group.

Hypothesis 3: The WAST© will have an inter-rater reliability of 70% (k=0.85).

DETAILED DESCRIPTION:
This study is a single-masked 2-centre randomized control trial. In order to evaluate the usability and feasibility of the app, we will evaluate 52 (26 female) patients and their physical therapists. Participants will be randomly assigned to either the experimental or control group, both of which will use apps available from Move Improve®. Through the Move Improve® platform, both groups will be shown instructional videos of different movement skills, and then will be able to record secure videos of themselves performing the skills. The control group will watch videos related to breathing skills and the treatment group will watch videos related to walking aids. Patients must be aged 18-80 years and require the regular (>75% of ambulatory time) use of a WA. Patients will be recruited from the South Health Campus Neuromuscular and Orthopedic Clinics, Foothills Medical Centre Orthopedic Surgery and Physiatry Clinics, Foothills Medical Centre Orthopedic Inpatients Units, Foothills Medical Centre Day Surgery Units, University of Calgary Sports Medicine Centre, Momentum Health Physiotherapy Clinics (all in Calgary, Alberta), and Centre interdisciplinaire de recherche en réadaptation et intégration sociale (CIRRIS, in Québec City, Québec) where they will be informed of the project during clinical sessions with their practitioners. Potential patient participants will be screened in-person by a Research Assistant to determine their eligibility.

The primary outcome of the study is the Activities-specific Balance Confidence (ABC) scale assessed at baseline and 4 weeks. Secondary outcomes include the following at baseline and 4 weeks: Timed Up and Go (TUG), 6-Minute Walk Test (6MWT), Berg Balance Score (BBS), Walking Aid Skills Test© (WAST©), number of falls, and a description of upper limb location and pain. Additionally, we will consider both the patient and clinician participant's perspectives about the perceived usefulness, ease of use of, and satisfaction with the app and will ask them about perceived treatment effect and additional time required during therapy sessions. Participant's time spent on and score of each component will also be recorded.

Eligible participants will sign consent forms to participate. During their usual physical therapy session, the patient will use the app on 2 occasions (up to 15 minutes). After the session, the patient will each be asked to complete online questionnaires via Qualtrics (Utah, USA) on the iPad. The questionnaires will include confidence using walking aid, comfort using walking aid, Activity-specific Balance Confidence (ABC) Scale, app ease of use, app usability, and app satisfaction. The Research Assistant will be available during the session in case problems arise.

A physical assessment will occur at baseline, 2-weeks, and 4-weeks after initial assessment. The physical assessment contains the BBS, 6MWT, and WAST©. This evaluation will be conducted by the Research Assistant.

The WAST© will be video recorded by the Research Assistant. We will ask physical therapists to rate the videos of the participants to determine the reliability and validity of the walking aid skills test.

There have been no published studies on the minimal clinically important difference of the ABC. A previous study on 376 knee osteoarthritis patients resulted in an increase in ABC scores by a mean of 9.15 at 1-year post-total knee arthroplasty. Using a repeated-measures Cohen's d, the effect size in that study was 0.585. As such, a sample size of 18 would be sufficient to explore two-tailed differences within a single individual over time on the ABC as they were recovering from their injury (1-β=0.8, α=0.05; G*Power, Germany). However, we would like to explore the differences between two groups (app exposures) as a primary outcome. We also wish to explore sex-based differences and want to incorporate a conservative estimate 10% dropout rate. As such, it is likely that 26 participants in each cohort will be sufficient to find significant differences for the primary outcome variable being investigated.

Participants will be randomly assigned to the experimental or control groups using 1:1 allocation ratio to increase the power to detect statistically significant differences between groups. To support balance between groups, a computerized randomization process, stratified by site (4 sites) and sex with block sizes of 2, 4, and 6, designed by a biostatician using SPSS3 (IBM, Armonk, USA) will be used.

Information on the baseline covariates will be presented for the two groups. Rates of non-participation will be reported. All primary and exploratory secondary mobility outcome measures will be assessed for normality using the Shapiro-Wilk test in SPSS (IBM, Armonk, USA). ABC scores will be analyzed using a two-way repeated measures analysis of variance with Greenhouse-Geisser correction with time and app group as factors. For the remaining variables, between-group differences will be investigated using either independent group t-tests or non-parametric Mann-Whitney U tests in SPSS. α = 0.05 will be used for all testing, with correction for multiple comparisons using the Benjamini-Hochberg approach.

Primary outcome variables will be analyzed in SPSS. Reliability will be analyzed in Microsoft Excel and will be investigated using independent and dependent group t-tests in Excel, with a p-value set at <0.05. Validity will be analyzed in Microsoft Excel and compared to predicted ability to walk, and the Walking Aid Skills Test scores compared to the Timed-Up and Go, Balance Scale and 2-minute Walk. Reliability will be analyzed in Microsoft Excel and compared scores of the same reviewer over time and between reviewers.

ELIGIBILITY:
Inclusion Criteria:

* patient at a study site currently using walking aids >75% of their ambulatory time
* age 18-99

Exclusion Criteria:

* currently using a wheelchair >25% of their ambulatory time
* cannot comfortably communicate in English or French
* history of significant cognitive or visual impairment that would affect their ability to use the app interventions
* unable to give voluntary informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Activities-specific Balance Confidence (ABC) | baseline, 2 weeks, 4 weeks
  16-item self-report measure that asks individuals to rate their balance confidence in performing a range of activities from 0% to 100%.

SECONDARY OUTCOMES:
2-minute walk test | baseline, 2 weeks, 4 weeks
  Measuring the distance walked in 2 minutes. The greater distance covered the more proficient participant is at using walking aid. Minimum: 0 metres. Maximum: unlimited.
Berg Balance Scale | baseline, 2 weeks, 4 weeks
  Scale ranges from 0 to 56. Higher score indicates better balance.
Timed Up and Go | baseline, 2 weeks, 4 weeks
  Patient will walk to a line that is 3m away from them, at the line they will turn around, walk 3m, and sit in a chair. The time stops when their buttocks touch the chair. A time of greater than or equal to 15 seconds indicates an increased fall risk.
Walking Aid Skills Test© | baseline, 2 weeks and 4 weeks
  Scale from 0-100 with higher value indicating greater proficiency using walking aid.

CONTACTS AND LOCATIONS:
Overall Officials: Ranita Manocha, MD, MSc, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - CIRRIS, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No
Anonymized IPD will be shared if requested on a case-by-case basis.

REFERENCES:
- [Background] Si HB, Zeng Y, Zhong J, Zhou ZK, Lu YR, Cheng JQ, Ning N, Shen B. The effect of primary total knee arthroplasty on the incidence of falls and balance-related functions in patients with osteoarthritis. Sci Rep. 2017 Nov 29;7(1):16583. doi: 10.1038/s41598-017-16867-4. PMID 29185496
- [Derived] Nindorera F, Manocha RHK, Miller WC, Routhier F, Best KL. Exploring the Influence of a Novel App for Training and Evaluating Walking Aid Skills in Walking Aid Users: Protocol for a Pragmatic Single-Blind Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 24;14:e71060. doi: 10.2196/71060. PMID 41442703